CLINICAL TRIAL: NCT04597281
Title: MEditerranean LIfestyle in Pediatric Obesity Prevention
Acronym: MELI-POP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Luis A. Moreno Aznar (Other)
Collaborators: Instituto Maimónides de Investigación Biomédica de Córdoba (Unknown); Fundación del Instituto de Investigación Sanitaria de Santiago (Unknown)
Responsible Party: Sponsor-Investigator, Luis A. Moreno Aznar, Professor, Universidad de Zaragoza
Organization: Universidad de Zaragoza (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: PI18/00666
Record Dates: First submitted 2020-09-28; First posted 2020-10-22 (Actual); Last update posted 2020-10-22 (Actual); Status verified 2020-10

CONDITIONS: Obesity, Childhood
MeSH Terms: conditions — Pediatric Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mediterranean lifestyle (Experimental): Mediterranean lifestyle, including dietary advice and physical activity advice. In addition, families receive extra-virgin olive oil and fish and two sessions of physical activity per week, for free.
  Interventions: Other: Lifestyle intervention
- Usual care (No Intervention): General care by their pediatricians.

INTERVENTIONS:
Other: Lifestyle intervention — The intervention group, will receive education on Mediterranean lifestyle (Mediterranean diet and physical activity promotion), combined with the provision of extra-virgin olive oil and fish, in order to be consumed at least 3 times per week. Physical activity sessions with a physical activity monitor will also be offered for free to the children (2 sessions of 60 minutes of moderate-vigorous physical activity, per week)
  Arms: Mediterranean lifestyle

SUMMARY:
The current project is a randomized controlled multi-centre clinical trial, in a cohort of children aged 3 to 6 years at baseline and being at obesity risk. The main objective consists on assessing the efficacy of an intervention during early childhood, considering a healthy lifestyle based on the promotion of a Mediterranean dietary pattern and regular physical activity, compared with a control group, on decreasing obesity incidence 5 and 10 years after the beginning of the intervention. It is envisaged to include 738 children, aged 3 to 6 years, having at baseline a body mass index (BMI) < than the equivalent to 30 kg/m2 in adults, and at least one parent having a BMI > 25 kg/m2. The clinical trial will have two arms and will be performed in Primary Health centres in 3 cities: Córdoba, Santiago de Compostela and Zaragoza. The control group will receive usual care by healthcare professionals. The intervention group, will receive education on Mediterranean lifestyle (Mediterranean diet and physical activity promotion), combined with the provision of extra-virgin olive oil and fish, in order to be consumed at least 3 times per week. Physical activity sessions with a physical activity monitor will also be offered for free to the children (2 sessions of 60 minutes of moderate-vigorous physical activity, per week). The participants' degree of compliance with the intervention will be periodically monitored. The main outcome is the incidence of obesity and the secondary outcomes are changes in body composition, physical fitness and cardiovascular risk factors. We are targeting for a 10 year follow-up.

DETAILED DESCRIPTION:
Hypothesis A healthy lifestyle, based on the promotion of the Mediterranean dietary pattern and regular physical activity, decrease the likelihood of developing obesity and cardio-metabolic abnormalities during childhood and adolescence.

Objectives

To assess, in a cohort of children at high risk of obesity, if an intervention during childhood and adolescence, considering a healthy lifestyle based on the promotion of Mediterranean dietary pattern and regular physical activity, when compared with a control group Main objective

1. To decrease obesity incidence 5 and 10 years after the start of the intervention Secondary objectives
2. To improve body composition (Body mass index z-score, Fat mass index z-score, waist circumference) assessed in a yearly basis
3. To improve health-related physical fitness assessed in a yearly basis
4. To improve cardiovascular risk factor (classic and omics) associated with obesity 1, 3, 5 and 10 years after the start of the intervention Intermediary objectives
5. To increase the adherence to a Mediterranean dietary pattern 1, 3, 5 and 10 years after the start of the intervention
6. To increase the adherence to age-specific physical activity recommendations 1, 3, 5 and 10 years after the start of the intervention

ELIGIBILITY:
Inclusion Criteria:

* Children > 3 years and < 7 years, with at least one parent having a BMI ≥ 25 kg/m2, with no disease responsible for the high BMI.
* Children with normal- or over weight, following the IOTF criteria (Cole TJ, Lobstein T. Pediatr Obes 2012; 7: 284-294).

Exclusion Criteria:

* Children < 3, or > 7 yearss, or both parents Having BMI <25 kg/m2.
* Children with chornic diseases or following a therapeutic diet .
* Children from families having dietary habits not fitting with the characteristics of the dietary intervention.
* Children from families having difficulties to follow the protocol.

Ages: 3 Years to 7 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 738 (Estimated)
Dates: Start 2018-03-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2032-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of obesity | 10 years
  Number of children having normal-weight at the baseline measurement and having obesity at follow-up.

SECONDARY OUTCOMES:
Body composition | 10 years
  Fat mass index assessed using skinfold thickness measurements.

CONTACTS AND LOCATIONS:
Overall Officials: Luis A Moreno Aznar, MD, PhD, Principal Investigator — Universidad de Zaragoza
Locations (3):
- Spain (3):
  - Instituto Maimónides de Investigación Biomédica de Córdoba, Córdoba
  - Fundación del Instituto de Investigación Sanitaria de Santiago, Santiago de Compostela
  - Instituto de Investigación Sanitaria Aragón, Zaragoza

IPD SHARING:
Plan to Share IPD: Yes
The plan is to allow other researchers to use the data obtained in the study is this is approved byut the corresponding responsible persons.
Supporting Information: Study Protocol, ICF, CSR, Analytic Code
Time Frame: At the end of the trial
Access Criteria: Approval of an analysis protocol by the study's steering committee

REFERENCES:
- [Derived] De Miguel-Etayo P, Flores-Rojas K, Vazquez-Cobela R, Jurado-Castro JM, Larruy-Garcia A, Picans-Leis R, Castro-Collado C, Pastor-Villaescusa B, Llorente-Cantarero FJ, Aguilera CM, Gil-Campos M, Leis R, Moreno LA; MELI-POP Study group. MELI-POP Study: MEditerranean LIfestyle in Pediatric Obesity Prevention. Study protocol for a randomized controlled trial. BMC Public Health. 2025 Nov 5;25(1):3791. doi: 10.1186/s12889-025-24351-2. PMID 41194137